CLINICAL TRIAL: NCT01003262
Title: Evaluating an Emergency Department Observation Syncope Protocol for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Southern California (Other); Brigham and Women's Hospital (Other); Corewell Health East (Other); Duke University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3163864; RC1AG035664-01 (NIH)
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Syncope
Keywords: Observation Unit; Emergency Department
MeSH Terms: conditions — Syncope; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Emergency Department Observation (Experimental): The EDOSP will consist of cardiac enzyme testing, 12-24 hours of cardiac monitoring, and echocardiogram testing by explicit criteria
  Interventions: Other: Emergency Department Observation Protocol
- Unstructured, inpatient evaluation (Active Comparator)
  Interventions: Other: Unstructured, inpatient evaluation

INTERVENTIONS:
Other: Emergency Department Observation Protocol — The EDOSP will consist of cardiac enzyme testing, 12-24 hours of cardiac monitoring, and echocardiogram testing by explicit criteria
  Arms: Emergency Department Observation
Other: Unstructured, inpatient evaluation — This is unstructured management by an inpatient medical team.
  Arms: Unstructured, inpatient evaluation

SUMMARY:
Syncope, defined as a transient loss of consciousness, accounts for over 700,000 annual U.S. emergency department visits and may herald a life-threatening condition in older adults (age≥60 years). Existing risk prediction instruments cannot reliably identify who among such older patients can safely be discharged home from an emergency department. As a result, the majority of older patients without a clear cause for syncope are hospitalized for diagnostic evaluation. However, current admission practices are characterized by low diagnostic yield, do not clearly improve outcomes, and account for over $2.4 billion in annual hospital costs. Most admitted patients are discharged within 48 hours, and approximately 50% of patients do not have an identified cause of syncope after their hospitalization.

The implementation of an expedited and standardized Emergency Department Observation Syncope Protocol (EDOSP) may safely reduce hospitalization of older patients with syncope. The investigators propose a pilot randomized trial to implement and evaluate EDOSP at two emergency departments. This study has the following exploratory Specific Aims:

1. To compare admission rates and length-of-stay associated with EDOSP to standard care.
2. To compare serious outcomes rates associated with EDOSP to standard care.
3. To compare quality-of-life associated with EDOSP to standard care.
4. To compare the incremental costs and cost-effectiveness of EDOSP to standard care.

Over a one-year period, 120 intermediate-risk older adults who present with syncope at the two study sites will be randomized to 1 of 2 arms: 1.) intervention arm: expedited and standardized EDOSP care; or 2.) control arm: routine care consisting of admission from the emergency department.

If this pilot trial suggests that EDOSP can safely reduce admissions, then the investigators will plan a larger study powered to evaluate clinical, quality-of-life, and economic outcomes. A successful EDOSP intervention would have important clinical policy implications and improve the emergency department care of older adults with syncope.

ELIGIBILITY:
Inclusion Criteria:

* Age≥60 years
* A complaint of syncope or near-syncope (Syncope is defined as a sudden, transient loss of consciousness. Near-syncope is defined as a sensation of imminent loss of consciousness, without actual syncope.)
* Intermediate risk of adverse outcome (see Table)
* Patient speaks either English or Spanish as a primary language.

Exclusion Criteria:

* Syncope mimics (intoxication, weakness or dizziness with syncope/ near-syncope, hypoglycemia, and cardiac arrest)
* New or baseline cognitive impairment or dementia)
* Inability to provide follow-up information (e.g. homeless or resides outside of U.S.)
* Inability to speak Spanish or English
* Low- and high-risk patients (see Table).

Risk Stratification Guidelines:

* High Risk
* Serious condition identified in ED
* History of ventricular arrhythmia
* Cardiac Device with dysfunction
* Presentation consistent with acute coronary ischemia

Intermediate Risk

* No High Risk features
* Presentation not consistent with orthostatic or vasovagal syncope

Low Risk

* Presentation consistent with orthostatic or vasovagal syncope

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Admission Rate | Enrollment date

SECONDARY OUTCOMES:
30 day clinical outcomes | 30 days
Quality of life | 30 days
Cost | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Sun, MD, MPP, Principal Investigator — University of California, Los Angeles
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oaks, Michigan
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Result] Sun BC, McCreath H, Liang LJ, Bohan S, Baugh C, Ragsdale L, Henderson SO, Clark C, Bastani A, Keeler E, An R, Mangione CM. Randomized clinical trial of an emergency department observation syncope protocol versus routine inpatient admission. Ann Emerg Med. 2014 Aug;64(2):167-75. doi: 10.1016/j.annemergmed.2013.10.029. Epub 2013 Nov 13. PMID 24239341